CLINICAL TRIAL: NCT05034094
Title: Auditory and Vestibular Functions in Patients With Parkinson's Disease
Brief Title: Auditory and Vestibular Function in Parkinson's Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Kamal Sabrah, resident, Assiut University
Other Study IDs: parkinson
Record Dates: First submitted 2021-08-09; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: VEMP recording — * Clinical evaluation: All participants will undergo detailed medical and neurological histories and examinations.
  * The severity of manifestations of PD will be assessed using the Movement Disorder Society (MDS)-sponsored new version of Unified PD Rating Scale (MDS-UPDRS).

SUMMARY:
The aims of this study are to:

1. Evaluate peripheral and central auditory and vestibular function in group of adults with idiopathic PD.
2. Determine the relationship between the presence of significant auditory and vestibular dysfunctions to patients' demographic, clinical (motor and non-motor manifestations) and treatment variables

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a progressive neurodegenerative disease of central nervous system that mainly affects the motor system . The worldwide data showed a rising prevalence of PD with age. Meta-analysis showed a prevalence of 41/100,000 in 40-49 years old; 107/100,000 in 50-59 years; 173/100,000 in 55-64 years; 428/10,000 in 60-69 years; 425/10,000 in 65-74 years; 1087/10,000 in 70-79 years; and 1903/100,000 in >80 years. Some differences in prevalence have been observed in different geographic location and in relation to sex . Patients with PD have multiple non-motor symptoms (NMSs) including fatigue, sensory symptoms, autonomic disturbance. sleep disorders, neuropsychiatric abnormalities etc . In the last decade and even in early stages of PD, studies reported hearing and/or vestibular dysfunctions in patients with PD with an estimated frequency of 25-50% . In the last decade and even in early stages of PD, studies reported vestibular dysfunctions in patients with PD with an estimated frequency of 14-25% compared to 5 -7.4% of the general population matched for age.

The pathophysiologic mechanisms of NMSs with PD are complex. Experimental as well as functional neuroimaging (e.g. SPECT and functional MRI) studies found that outputs from basal ganglia are directed to the inferior colliculus, medial geniculate nucleus, and temporal cortex. Motor or NMSs, occur due to loss not only of dopaminergic neurons in the substantia nigra but also in other dopaminergic and non-dopaminergic areas of the brain including serotoninergic, noradrenergic, and cholinergic systems. Lewy bodies and neurites consisting of α-synuclein, the main pathological features of PD, were observed in brain hemispheres as well as, spinal cord, brainstem nuclei and fiber tracts including vestibular nuclei and efferent neuronal system within the inner ear .

Diagnostic basic audiologic and vestibular evaluation and electrophysiological testing as brainstem auditory evoked potential (BAEP), videonystagmography (VNG) and cervical (cVEMP) and ocular (oVEMP) vestibular evoked myogenic potentials are easily available and applicable in many parts of the world as diagnostic tests to objectively evaluate peripheral and central auditory and vestibular dysfunctions for many disease including PD . This may provide early drug intervention and rehabilitation for patients and improve their qualities of life.

ELIGIBILITY:
Inclusion Criteria:

* Adults with age range 55-65 years old from both gender.
* Patients have to fulfil the criteria for diagnosis of idiopathic PD [Postuma et al., 2015]. and age, sex and socioeconomic matched healthy subjects recruited from the general population as controls for statistical comparisons.

Exclusion Criteria:

* - Concomitant medical and metabolic illnesses.
* Secondary or atypical parkinsonism
* Evidence of concomitant cerebrovascular stroke temporally related to the onset of the disease.
* Major psychiatric disorder known to affect cognition.
* Dementia (i.e. mini mental score examination or MMSE score <24)
* Major language disturbance
* MRI brain showing structural lesion
* Severe known auditory (hearing thresholds >50 dBnHL) or visual impairment affecting their ability to complete testing before participation of the study.
* Improper neck movements that interfere with assessment.
* Middle ear diseases, ear infection, ear trauma, or acoustic trauma

Ages: 55 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — old age
Study Population: * Patients with PD will be recruited from the Department of Neurology and Psychiatry and its out-patient clinic, Assiut University Hospital, Assiut, Egypt.
  * All patients will be encoded to confidentiality.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-08-13 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Auditory and vestibular functions in patients with Parkinson's disease | 16 month
  1.1 basic audiological evaluation this include otoscopic examination , screening audiogram,stapedial reflex testing 1.2 vestibular evaluation by VNG recording ,VEMP recording ,cVEMP recording ,oVEMP recording

REFERENCES:
- [Background] Smith PF. Vestibular Functions and Parkinson's Disease. Front Neurol. 2018 Dec 11;9:1085. doi: 10.3389/fneur.2018.01085. eCollection 2018. PMID 30619045
- [Background] Scarpa A, Cassandro C, Vitale C, Ralli M, Policastro A, Barone P, Cassandro E, Pellecchia MT. A comparison of auditory and vestibular dysfunction in Parkinson's disease and Multiple System Atrophy. Parkinsonism Relat Disord. 2020 Feb;71:51-57. doi: 10.1016/j.parkreldis.2020.01.018. Epub 2020 Jan 30. PMID 32032926